CLINICAL TRIAL: NCT05774171
Title: To Explore the Protective Effect of SARS-CoV-2 Vaccination on Cancer Patients Infected With SARS-CoV-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: SH-2022018
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Infection; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples were collected from cancer patients who had been infected with SARS-CoV-2, with or without previous SARS-CoV-2 vaccination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients with SARS-CoV-2 vaccination: Cancer patients with SARS-CoV-2 vaccination
  Interventions: Other: no intervention
- Cancer patients without SARS-CoV-2 vaccination: Cancer patients without SARS-CoV-2 vaccination
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
For tumor patients, the virus antibody titer produced by the SARS-CoV-2 vaccine is often lower than that of normal people in a short period of time, but in the long run, it can significantly reduce the infection rate and fatality rate of the new coronavirus, and the adverse reactions are mild and there is no significant difference with normal people. However, there is still no real-world research data in China to prove the protective effect of the SARS-CoV-2 vaccine on patients with tumors infected with the SARS-CoV-2 virus.

DETAILED DESCRIPTION:
To explore the protective effect of SARS-CoV-2 vaccination on cancer patients infected with SARS-CoV-2. Serum samples were collected from cancer patients who had been infected with SARS-CoV-2 and were previously vaccinated or unvaccinated. The SARS-CoV-2 antibodies (IgG and IgM concentrations) were detected by micro-magnetic particle chemiluminescence method, and the differences were compared. The results of this real-world prospective cohort study can be used to guide the vaccination of cancer patients in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years old, regardless of gender;
2. patients with previous or current tumor, regardless of tumor type;
3. have a history or current infection with SARS-CoV-2;
4. The vital signs were stable, without severe pulmonary, heart, liver and other important organ dysfunction;
5. those with good compliance, agreed to participate in this clinical study, receive corresponding treatment, and signed the informed consent.

Exclusion Criteria:

1. Those who do not meet the inclusion criteria or diagnostic criteria, and cannot cooperate with blood sampling and arrangement;
2. patients with severe bleeding disorders such as coagulopathy or essential thrombocytopenia;
3. local skin ulceration affecting blood drawing, severe rash, or infectious diseases;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. age > 18 years old, regardless of gender;
  2. patients with previous or current tumor, regardless of tumor type;
  3. have a history or current infection with SARS-CoV-2;
  4. The vital signs were stable, without severe pulmonary, heart, liver and other important organ dysfunction;
  5. those with good compliance, agreed to participate in this clinical study, receive corresponding treatment, and signed the informed consent.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of SARS-CoV-2 antibodies of all patients | 2022.12-2022.6 Clear experimental scheme;Serum antibody detection and data collection were completed 2022.7-2022.8 The follow-up data analysis was completed 2022.8-2022.9 Conduct the writing and submission of the paper
  Detection of SARS-CoV-2 antibodies (IgG and IgM concentrations) by micro-magnetic particle chemiluminescence method of all patients

CONTACTS AND LOCATIONS:
Overall Officials: yuan peng, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Sanhuan Cancer Hospital, Chaoyang District, Beijing(Cancer Hospital, Chinese Academy of Medical Sciences, close medical alliance), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirsch C, Zorger AM, Baumann M, Park YS, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with solid tumours. Cochrane Database Syst Rev. 2025 Apr 16;4(4):CD015551. doi: 10.1002/14651858.CD015551.pub2. PMID 40237463